CLINICAL TRIAL: NCT02320240
Title: Serotonin-norepinephrine Reuptake Inhibitors and Acute Kidney Injury
Acronym: SNRI-AKI
Status: Completed | Type: Observational
Sponsor: Canadian Network for Observational Drug Effect Studies, CNODES (Other)
Collaborators: Drug Safety and Effectiveness Network, Canada (Other); Canadian Institutes of Health Research (CIHR) (Other Government)
Responsible Party: Sponsor
Other Study IDs: Q12-08
Record Dates: First submitted 2014-12-16; First posted 2014-12-19 (Estimated); Last update posted 2016-03-14 (Estimated); Status verified 2016-03

CONDITIONS: Depression; Acute Kidney Injury
Keywords: antidepressants; acute kidney injury; SNRI; renal failure; duloxetine; CNODES
MeSH Terms: conditions — Depression; Acute Kidney Injury; Renal Insufficiency | interventions — Duloxetine Hydrochloride; Venlafaxine Hydrochloride; Desvenlafaxine Succinate; Citalopram; Escitalopram; Fluoxetine; Fluvoxamine; Paroxetine; Sertraline

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- SNRI Exposure Group: Patients who received a new prescription for an SNRI (duloxetine, venlafaxine, or desvenlafaxine at any dosage) with no prescriptions for either SNRI or SSRI in the prior year.
  Interventions: Drug: Duloxetine; Drug: Venlafaxine; Drug: Desvenlafaxine
- SSRI Exposure Group: Patients who received a new prescription for an SSRI (citalopram, escitalopram, fluoxetine, fluvoxamine, paroxetine, or sertraline at any dosage) with no prescriptions for either SSRI or SNRI in the prior year.
  Interventions: Drug: Citalopram; Drug: Escitalopram; Drug: Fluoxetine; Drug: Fluvoxamine; Drug: Paroxetine; Drug: Sertraline

INTERVENTIONS:
Drug: Duloxetine — Current exposure to Duloxetine will be defined as a prescription lasting until the index date or dispensed in the 60 days before the index date.
  Groups: SNRI Exposure Group
Drug: Venlafaxine — Current exposure to Venlafaxine will be defined as a prescription lasting until the index date or dispensed in the 60 days before the index date.
  Groups: SNRI Exposure Group
Drug: Desvenlafaxine — Current exposure to Desvenlafaxine will be defined as a prescription lasting until the index date or dispensed in the 60 days before the index date.
  Groups: SNRI Exposure Group
Drug: Citalopram — Current exposure to Citalopram will be defined as a prescription lasting until the index date or dispensed in the 60 days before the index date.
  Groups: SSRI Exposure Group
Drug: Escitalopram — Current exposure to Escitalopram will be defined as a prescription lasting until the index date or dispensed in the 60 days before the index date.
  Groups: SSRI Exposure Group
Drug: Fluoxetine — Current exposure to Fluoxetine will be defined as a prescription lasting until the index date or dispensed in the 60 days before the index date.
  Groups: SSRI Exposure Group
Drug: Fluvoxamine — Current exposure to Fluvoxamine will be defined as a prescription lasting until the index date or dispensed in the 60 days before the index date.
  Groups: SSRI Exposure Group
Drug: Paroxetine — Current exposure to Paroxetine will be defined as a prescription lasting until the index date or dispensed in the 60 days before the index date.
  Groups: SSRI Exposure Group
Drug: Sertraline — Current exposure to Sertraline will be defined as a prescription lasting until the index date or dispensed in the 60 days before the index date.
  Groups: SSRI Exposure Group

SUMMARY:
The purpose of this study is to determine if there is an excess risk of acute kidney injury (AKI) with Serotonin-norepinephrine reuptake inhibitors (SNRIs) as compared to Selective serotonin reuptake inhibitors (SSRIs), two classes of medication used for the treatment of depression.

DETAILED DESCRIPTION:
We plan to conduct retrospective population-based cohort studies within eight administrative databases from Canada, the United States, and the United Kingdom. Within each cohort, a nested case-control analysis will be performed to estimate incidence rate ratios (RR) of AKI associated with SNRIs compared to SSRIs using conditional logistic regression, with adjustment for high-dimensional propensity scores at baseline. The overall effect across sites will then be estimated using meta-analytic methods.

ELIGIBILITY:
Inclusion Criteria:

* A first prescription of an antidepressant of the SNRI or SSRI class of any dose between January 1, 1997 and March 31, 2010.

Exclusion Criteria:

* They were <12 years old at the time of cohort entry.
* They had less than 1 year of information in the database prior to the date of cohort entry.
* They had a prescription of an SNRI or SSRI in the year before the date of cohort entry.
* They had a prescription for both an SNRI and an SSRI on the day of cohort entry.
* They had a history of chronic kidney disease (including kidney transplantation and dialysis) or AKI in the year preceding cohort entry.
* The subject was previously included in the cohort.

Min Age: 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: The cohort will be formed of all patients in the databases aged 12 or older (or 65 or older in some of the databases) with a first prescription of an antidepressant of the SNRI or SSRI class of any dose between January 1, 1997 and March 31, 2010. The databases to be included are eight administrative databases from Canada (Alberta, Manitoba, Nova Scotia, Ontario, Quebec, and Saskatchewan), the United States (US MarketScan), and the United Kingdom (CPRD).
Sampling Method: Probability Sample
Enrollment: 3255526 (Actual)
Dates: Start 2013-06; Primary Completion 2014-12 (Actual); Study Completion 2014-12 (Actual)

PRIMARY OUTCOMES:
Acute Kidney Injury (AKI) | 2 years
  AKI will be defined as patients hospitalized with one of the following diagnosis codes for AKI in any of the listed diagnoses: ICD-9-CM codes 584, 584.5, 584.6, 584.7, 584.8, or 584.9; ICD-10 N17, N17.0, N17.1, N17.2, N17.8, or N17.9.

CONTACTS AND LOCATIONS:
Overall Officials: Pierre Ernst, MD, MSc, Principal Investigator — Lady Davis Institute for Medical Research, Jewish General Hospital - McGill University
Locations (1):
- Lady Davis Institute for Medical Research, Jewish General Hospital, Montreal, Quebec, Canada

REFERENCES:
- [Result] Renoux C, Lix LM, Patenaude V, Bresee LC, Paterson JM, Lafrance JP, Tamim H, Mahmud SM, Alsabbagh MW, Hemmelgarn B, Dormuth CR, Ernst P; Canadian Network of Observational Drug Effect Studies (CNODES) Investigators. Serotonin-Norepinephrine Reuptake Inhibitors and the Risk of AKI: A Cohort Study of Eight Administrative Databases and Meta-Analysis. Clin J Am Soc Nephrol. 2015 Oct 7;10(10):1716-22. doi: 10.2215/CJN.11271114. Epub 2015 Jul 31. PMID 26231193
- See also: This organization's website describing general functions, other CNODES projects, and investigator profiles. — http://www.cnodes.ca